CLINICAL TRIAL: NCT02118077
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Group Sequential Trial of G17DT for the Treatment of Advanced Pancreatic Cancer.
Brief Title: Sequential Trial of G17DT for the Treatment of Advanced Pancreatic Cancer
Acronym: PC6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC6
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- G17DT (Experimental): 250 µg administered at Weeks 0,1,3 and 24 by intramuscular injection, followed by additional injections (boosters) of 250 µg every 6 months at investigator's discretion.
  Interventions: Biological: G17DT
- Placebo (Placebo Comparator): Placebo administered at Weeks 0, 1, 3, and 24 by intramuscular injection followed by additonal injections of placebo every 6 months.

INTERVENTIONS:
Biological: G17DT
  Arms: G17DT

SUMMARY:
Compare the effect of G17DT with that of placebo on the survival of subjects with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a histologically or cytologically confirmed diagnosis of pancreatic carcinoma, who were not eligible for tumor resection with curative intent (i.e., Stage II, III, or IV disease)
* Male or female subjects over 18 years of age
* Subjects with a life expectancy of at least 2 months
* KPS score of ≥60%
* Written informed consent

Exclusion Criteria:

* Previous, concomitant, or anticipated use (up to Week 12) of chemotherapy, radiotherapy, immunotherapy, or any other anticancer therapy
* Previous (during the 4 weeks before the study), concomitant, or anticipated use (up to Week 12) of immunosuppressants. However, for systemic [i.e., oral or injected] corticosteroids, previous use and concomitant use at study entry were prohibited, while introduction during the course of the study was permitted.)
* History of other malignant tumor within the previous 5 years, except nonmelanomatous skin cancer, and in situ carcinoma of the uterine cervix
* Known immunodeficiency
* Females who were pregnant, planning to become pregnant, or lactating (Women who, in the opinion of the investigator, were of childbearing potential were to have a negative pregnancy test before study drug administration.)
* Subjects taking part in another study involving an investigational or licensed drug or device in the 3 months preceding enrollment or up to Week 12 during this study
* Previous G17DT treatment
* Hematological indicators as follows:

  * Hemoglobin <9.5 g/dL
  * Neutrophils <2.0 × 109/L
  * Platelets <100 × 109/L
* Any other condition or circumstance that might have the following results:

  * Worsen if the subject participated in the study
  * Reduce the subject's ability to comply with the protocol
  * Confound the interpretation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2001-04; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Patient Survival | Up to week 134
  The vital status of each patient was followed until death or end of the study.
Number of Participants with Serious and Non-Serious Adverse Events | up to week 134
  Adverse events, defined as any event involving adverse reactions, illnesses with onset during the study, or exacerbations of pre-exisiting illnesses, were assessed at each visit.

SECONDARY OUTCOMES:
Objective tumor response | Weeks 24 and 52
  Patients were monitored for an objective tumor response measured by means of an abdomincal computed tomography.